CLINICAL TRIAL: NCT00543738
Title: MK0767 and Metformin Combination Study (0767-028)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-028; 2007_639; MK-0767-028
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
A study to test the effects of MK0767 when added to Metformin in patients with inadequately controlled Type 2 Diabetes Mellitus.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* All women of childbearing potential must have a negative urine pregnancy test prior to starting the study
* Patients must be on a stable dose of metformin for at least 2 weeks prior to visit 2

Exclusion Criteria:

* Patients with a history of type 1 diabetes mellitus and/or history of ketoacidosis
* Patients on estrogen replacement therapy regimen or SERM
* Patients with history of, allergy to, intolerance or hypersensitivity to statins or fibric acid derivatives, including history of elevated muscle and liver function tests, jaundice, hepatoxicity, or myopathy associated with these treatments
* Patient is on a weight loss program with ongoing weight loss or starting an intensive exercise program within 4 weeks from starting the study
* Have active liver or gall bladder disease
* HIV positive

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2003-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC